CLINICAL TRIAL: NCT02421406
Title: An Internet-based Behavioral Weight Loss Program for HIV+ Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2P30AI042853-16 (NIH); P30AI042853 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-04-20 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-01

CONDITIONS: Overweight; Obesity; HIV
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Behavioral Intervention (Experimental): Participants receive a 12-week Internet-based eating and activity intervention including multimedia lessons and enhanced self-monitoring of weight loss behaviors with automated feedback
  Interventions: Behavioral: Internet Behavioral Intervention
- Internet Education Intervention (Active Comparator): Participants receive 12 weekly Internet-based weight loss lessons containing information for modification of diet and activity behaviors, but not behavioral strategies for changing these behaviors.
  Interventions: Behavioral: Internet Education Intervention

INTERVENTIONS:
Behavioral: Internet Behavioral Intervention — A series of 12 multi-media lessons will be accessible to participants on their own computers. The lessons (each of which takes about 15 minutes to complete) are based on the Diabetes Prevention Program (DPP) and Look AHEAD. Participants will be taught to record their weight, the calories and the fat grams in each food item, and their physical activity (in minutes) on a daily basis. At the end of the week, they will submit their self-monitored information to the study website and receive an automated feedback message about their progress to date. The lessons will also present key behavior change strategies such as cognitive restructuring, problem solving and relapse prevention.
  Arms: Internet Behavioral Intervention
Behavioral: Internet Education Intervention — A series of 12 lessons will be accessible to participants on their own computers. Participants will be given information about normal, overweight and obese categories of body mass index, and provided information on the health problems that are associated with being overweight and the benefits of weight loss for treating and preventing such problems. General information about healthy eating will be provided. Participants will be educated about the benefits of increasing their physical activity, and strategies for increasing activity safely.
  Arms: Internet Education Intervention

SUMMARY:
The goal of this project is to determine whether an Internet-based weight loss program will lead to weight loss and improvements in cardiovascular disease risk factors in people living with HIV.

DETAILED DESCRIPTION:
The goal of this project is to provide an empirically validated weight loss program to HIV+ patients and evaluate its efficacy for weight loss and improvements in cardiovascular disease risk factors. Investigators will conduct a randomized pilot study with 50 overweight or obese patients who are HIV+, are recruited from the Miriam Hospital Immunology Center, and are interested in losing weight. These patients will be randomly assigned to a 12 week behavioral weight loss program delivered via the Internet or to a 12 week education only control group (also Internet based). Primary aims of this study are 1) to determine whether an Internet program is appropriate for this patient population, assessed by the success of recruiting 50 patients for the trial and their level of adherence over the 12 weeks, 2) to compare weight losses at the end of the 12 week program for program for patients randomized to the Internet behavioral weight reduction program (WT LOSS) relative to the Internet education program (CONTROL), 3) to compare the efficacy of the WT LOSS program relative to CONTROL for improving lipids (total cholesterol, HDL, LDL, triglycerides), metabolic measures (fasting blood sugar, insulin), and inflammatory markers (IL-6, C-reactive protein, adiponectin), and 4) to compare the changes in dietary intake and physical activity from baseline to 12 weeks in the WT LOSS and CONTROL conditions. Investigators will also store blood for later analysis of other adipokines (leptin) and biomarkers of microbial gut translocation (e.g., sCD14). These will provide important pilot data for future NIH funding related to both the implementation of weight loss programs and the effect of weight loss on the co-morbidities in this population.

ELIGIBILITY:
Inclusion Criteria:

* Recruited from the Miriam Hospital Immunology Center
* HIV+ with a CD4 count >200 and an undetectable viral load
* BMI greater than 27 kg/m2
* No health problems that make weight loss or unsupervised exercise unsafe
* English speaking
* Have access to a computer and the Internet

Exclusion Criteria:

* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Active substance abuser
* Currently pregnant or intend to become pregnant in the next 6 months
* Planning to move outside of the state within the next 6 months
* Have participated in a study conducted by the Weight Control & Diabetes Research Center in the past 2 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Weight | 12 weeks

SECONDARY OUTCOMES:
Diet assessed by 24-hour recalls | 12 weeks
  Dietary intake patterns measured using a three-day diet record.
Physical activity assessed by objective monitoring of activity | 12 weeks
  Objective physical activity measured using SenseWear Mini armband and self-reported physical activity measured using the International Physical Activity Questionnaire short form.
Metabolic profile assessed by analysis of fasting blood work | 12 weeks
  Fasting blood sugar and insulin measured using blood samples taken in fasting state.
Lipid profile assessed by analysis of fasting blood work | 12 weeks
  Lipids (total cholesterol, HDL, LDL, triglycerides) measured using blood samples taken in fasting state.
Inflammatory profile assessed by analysis of fasting blood work | 12 weeks
  IL-6, C-reactive protein, adiponectin measured using blood samples taken in fasting state.

REFERENCES:
- [Derived] Wing RR, Becofsky K, Wing EJ, McCaffery J, Boudreau M, Evans EW, Unick J. Behavioral and Cardiovascular Effects of a Behavioral Weight Loss Program for People Living with HIV. AIDS Behav. 2020 Apr;24(4):1032-1041. doi: 10.1007/s10461-019-02503-x. PMID 31004243
- [Derived] Becofsky K, Wing EJ, McCaffery J, Boudreau M, Wing RR. A Randomized Controlled Trial of a Behavioral Weight Loss Program for Human Immunodeficiency Virus-Infected Patients. Clin Infect Dis. 2017 Jul 1;65(1):154-157. doi: 10.1093/cid/cix238. PMID 28369269